CLINICAL TRIAL: NCT00635219
Title: A Randomised, Double-blind, Parallel-group, Placebo-controlled, Duloxetine-referenced, Fixed-dose Study Evaluating the Efficacy and Safety of Three Dosages of [Vortioxetine] Lu AA21004, in Acute Treatment of Major Depressive Disorder
Brief Title: Randomised Placebo-controlled Duloxetine-referenced Efficacy and Safety Study of 2.5, 5 and 10 mg of Vortioxetine (Lu AA21004) in Acute Treatment of Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 11984A; EudraCT 2007-001870-95 (Registry Identifier: EudraCT)
Record Dates: First submitted 2008-03-03; First posted 2008-03-13 (Estimated); Results first posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2013-12

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; Placebo-controlled; Active reference; Multicenter study; Randomised study; Acute treatment
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Vortioxetine: 2.5 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Vortioxetine: 5 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Vortioxetine: 10 mg (Experimental)
  Interventions: Drug: Vortioxetine (Lu AA21004)
- Duloxetine: 60 mg (Other): Active reference
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Placebo — capsules; daily; orally
  Arms: Placebo
Drug: Vortioxetine (Lu AA21004) — 2.5 mg/day; encapsulated tablets; orally
  Other Names: Brintellix
  Arms: Vortioxetine: 2.5 mg
Drug: Vortioxetine (Lu AA21004) — 5 mg/day; encapsulated tablets; orally
  Other Names: Brintellix
  Arms: Vortioxetine: 5 mg
Drug: Vortioxetine (Lu AA21004) — 10 mg/day; encapsulated tablets; orally
  Other Names: Brintellix
  Arms: Vortioxetine: 10 mg
Drug: Duloxetine — 60 mg/day; encapsulated capsules; orally
  Other Names: Cymbalta®
  Arms: Duloxetine: 60 mg

SUMMARY:
The purpose of the study is to evaluate the efficacy and the tolerability of three fixed doses of Vortioxetine in order to establish the appropriate clinical effective dose range in the treatment of Major Depressive Disorder (MDD).

ELIGIBILITY:
Inclusion Criteria:

* MDE as primary diagnosis according to DSM-IV-TR criteria (classification code 296.xx)
* Moderate to severe depression
* Current MDE duration of at least 3 months

Exclusion Criteria:

* Any current psychiatric disorder other than MDD as defined in the DSM-IV TR
* Any substance disorder within the previous 6 months
* Female patients of childbearing potential who are not using effective contraception
* Use of any psychoactive medication 2 weeks prior to screening and during the study

Other protocol-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 766 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com

REFERENCES:
- [Result] Baldwin DS, Loft H, Dragheim M. A randomised, double-blind, placebo controlled, duloxetine-referenced, fixed-dose study of three dosages of Lu AA21004 in acute treatment of major depressive disorder (MDD). Eur Neuropsychopharmacol. 2012 Jul;22(7):482-91. doi: 10.1016/j.euroneuro.2011.11.008. Epub 2011 Dec 30. PMID 22209361
- [Derived] Belzeaux R, Gorgievski V, Fiori LM, Lopez JP, Grenier J, Lin R, Nagy C, Ibrahim EC, Gascon E, Courtet P, Richard-Devantoy S, Berlim M, Chachamovich E, Theroux JF, Dumas S, Giros B, Rotzinger S, Soares CN, Foster JA, Mechawar N, Tall GG, Tzavara ET, Kennedy SH, Turecki G. GPR56/ADGRG1 is associated with response to antidepressant treatment. Nat Commun. 2020 Apr 2;11(1):1635. doi: 10.1038/s41467-020-15423-5. PMID 32242018
- [Derived] Christensen MC, Florea I, Loft H, McIntyre RS. Efficacy of vortioxetine in patients with major depressive disorder reporting childhood or recent trauma. J Affect Disord. 2020 Feb 15;263:258-266. doi: 10.1016/j.jad.2019.11.074. Epub 2019 Nov 13. PMID 31818787
- [Derived] Belzeaux R, Fiori LM, Lopez JP, Boucekine M, Boyer L, Blier P, Farzan F, Frey BN, Giacobbe P, Lam RW, Leri F, MacQueen GM, Milev R, Muller DJ, Parikh SV, Rotzinger S, Soares CN, Uher R, Foster JA, Kennedy SH, Turecki G. Predicting Worsening Suicidal Ideation With Clinical Features and Peripheral Expression of Messenger RNA and MicroRNA During Antidepressant Treatment. J Clin Psychiatry. 2019 May 7;80(3):18m12556. doi: 10.4088/JCP.18m12556. PMID 31087825
- [Derived] McIntyre RS, Florea I, Tonnoir B, Loft H, Lam RW, Christensen MC. Efficacy of Vortioxetine on Cognitive Functioning in Working Patients With Major Depressive Disorder. J Clin Psychiatry. 2017 Jan;78(1):115-121. doi: 10.4088/JCP.16m10744. PMID 27780334

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The patients were recruited from psychiatric settings.
Pre-assignment Details: The study consisted of a Screening Period; an 8-week Core Treatment Period; a 1-week double-blind downtaper period (Week 9); and a 4-week Safety Follow-up Period - the 4-week period after completion/withdrawal (Weeks 9 to 12).
Groups:
- Vortioxetine 2.5 mg; Vortioxetine 5 mg; Vortioxetine 10 mg: encapsulated tablets; orally
- Duloxetine 60 mg: encapsulated capsules; orally
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Started | 148 | 155 | 157 | 151 | 155
Completed | 123 | 130 | 122 | 117 | 113
Not Completed | 25 | 25 | 35 | 34 | 42
Not completed — Adverse Event | 12 | 10 | 18 | 15 | 19
Not completed — Lack of Efficacy | 5 | 6 | 3 | 4 | 6
Not completed — Non-compliance With Study Product | 0 | 0 | 0 | 2 | 1
Not completed — Protocol Violation | 0 | 2 | 3 | 2 | 4
Not completed — Withdrawal of Consent | 8 | 6 | 8 | 11 | 8
Not completed — Lost to Follow-up | 0 | 0 | 2 | 0 | 3
Not completed — Administrative or Other Reasons | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full-analysis set (FAS) - all patients in the all-patients-treated set (APTS) who had at least one valid postbaseline assessment of the primary efficacy variable
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 148 | 155 | 157 | 151 | 155 | 766
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.4 (12.5) | 46.0 (12.5) | 44.7 (13.1) | 45.2 (13.1) | 45.3 (12.0) | 44.9 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 110 | 104 | 100 | 105 | 522
  Male | 45 | 45 | 53 | 51 | 50 | 244
MADRS [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
  units on a scale | 31.7 (4.3) | 31.6 (4.0) | 32.7 (4.8) | 31.8 (3.9) | 31.4 (4.2) | 31.9 (4.3)
HAM-D-24 [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
  units on a scale | 29.8 (5.1) | 29.6 (5.8) | 31.3 (5.8) | 30.4 (5.4) | 29.9 (5.8) | 30.2 (5.6)
CGI-S [Mean (Standard Deviation); unit: units on a scale] — The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
  units on a scale | 4.8 (0.7) | 4.8 (0.7) | 4.8 (0.7) | 4.7 (0.7) | 4.7 (0.7) | 4.8 (0.7)
SDS [Mean (Standard Deviation); unit: units on a scale] — The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
  units on a scale | 19.9 (5.8) | 19.4 (6.5) | 19.6 (6.2) | 19.6 (6.5) | 19.2 (5.9) | 19.6 (6.2)
HAM-A [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
  units on a scale | 23.1 (5.6) | 22.2 (6.7) | 23.5 (6.2) | 23.4 (6.3) | 22.8 (6.4) | 23.0 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in MADRS Total Score After 8 Weeks of Treatment
Description: The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 (no symptom) to 6 (severe symptom). The 10 items represent the core symptoms of depressive illness. The rating should be based on a clinical interview with the patient, moving from broadly phrased questions about symptoms to more detailed ones, which allow a precise rating of severity, covering the last 7 days. Total score from 0 to 60. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: Full-analysis set (FAS) - all patients in the all-patients-treated set (APTS) who had at least one valid post-baseline assessment of the primary efficacy variable; last observation carried forward (LOCF); analysis of covariance (ANCOVA)
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 155 | 151 | 149
units on a scale | -14.8 (0.82) | -16.2 (0.79) | -16.5 (0.80) | -16.3 (0.80) | -16.8 (0.81)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; As soon as an endpoint was non-significant at the 0.025 level of significance, the testing procedure was stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.1321, ANCOVA — Since p-value >0.025, hierarchically testing stopped here; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-3.92 to 0.51], Standard Error of Mean 1.13 — To adjust for multiplicity the two doses of vortioxetine were tested separately versus placebo in the primary and key secondary efficacy analyses at a Bonferroni-corrected significance level of 0.025
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1847, ANCOVA — Since p-value >0.025, hierarchically testing stopped here; Mean Difference (Final Values) = -1.50, 95% CI 2-sided [-3.73 to 0.72], Standard Error of Mean 1.13 — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.2187, ANCOVA — This dose was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -1.38, 95% CI 2-sided [-3.59 to 0.82], Standard Error of Mean 1.12
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0741, ANCOVA — This treatment arm was not in the testing sequence. A nominal p-value is provided; Mean Difference (Final Values) = -2.04, 95% CI 2-sided [-4.27 to 0.20], Standard Error of Mean 1.14

2. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 8 Weeks of Treatment
Description: The Hamilton Depression Scale - 24 Items (HAM-D-24) measures depression severity. Items are rated on a scale from 0 (symptoms not present) to a maximum of 2 to 4 (symptom extremely severe) for a total score range of 0 to 76. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 155 | 151 | 149
units on a scale | -13.3 (0.82) | -14.4 (0.79) | -15.0 (0.80) | -14.9 (0.80) | -15.7 (0.81)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.1120, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.79, 95% CI 2-sided [-4.01 to 0.42], Standard Error of Mean 1.13 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.1487, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.63, 95% CI 2-sided [-3.85 to 0.59], Standard Error of Mean 1.13 — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.3246, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.11, 95% CI 2-sided [-3.31 to 1.10], Standard Error of Mean 1.12 — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0298, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -2.47, 95% CI 2-sided [-4.70 to -0.24], Standard Error of Mean 1.13 — No correction for multiplicity was made

3. Secondary Outcome: Proportion of Responders at Week 8 (Response Defined as a >=50% Decrease in the MADRS Total Score From Baseline)
Time Frame: Week 8
Population: FAS; LOCF; Logistic Regression
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 155 | 151 | 149
percentage of patients | 46.9 | 54.2 | 56.1 | 57.6 | 57.1
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.1370, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.90 to 2.23] — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0664, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.97 to 2.43] — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.2023, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.85 to 2.12] — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0765, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 1.52, 95% CI 2-sided [0.96 to 2.40] — No correction for multiplicity was made

4. Secondary Outcome: Change in Clinical Status Using CGI-I Score at Week 8
Description: The Clinical Global Impression - Global Improvement (CGI-I) is a 7-point scale rated from 1 (very much improved) to 7 (very much worse). The investigator rated the patient's overall improvement relative to baseline, whether or not, in the opinion of the investigator, this was entirely due to the drug treatment.
Time Frame: Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 154 | 151 | 149
units on a scale | 2.52 (0.10) | 2.32 (0.10) | 2.32 (0.10) | 2.35 (0.10) | 2.31 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.1436, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.47 to 0.07], Standard Error of Mean 0.14 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.2114, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.44 to 0.10], Standard Error of Mean 0.14 — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.1389, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.47 to 0.07], Standard Error of Mean 0.14 — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.1271, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.48 to 0.06], Standard Error of Mean 0.14 — No correction for multiplicity was made

5. Secondary Outcome: Change From Baseline in HAM-D-24 Total Score After 8 Weeks of Treatment in Patients With Baseline HAM-A Total Score >=20
Time Frame: Baseline and Week 8
Population: Patients With Baseline HAM-A Total Score >=20: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 97 | 91 | 100 | 101 | 92
units on a scale | -14.7 (1.10) | -14.3 (1.15) | -15.8 (1.09) | -15.8 (1.07) | -17.3 (1.14)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.4421, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-4.08 to 1.79], Standard Error of Mean 1.49 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.4399, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.15, 95% CI 2-sided [-4.07 to 1.77], Standard Error of Mean 1.49 — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.8093, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = 0.37, 95% CI 2-sided [-2.65 to 3.40], Standard Error of Mean 1.54 — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0897, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -2.60, 95% CI 2-sided [-5.61 to 0.41], Standard Error of Mean 1.53 — No correction for multiplicity was made

6. Secondary Outcome: Change From Baseline in SDS Total Score After 8 Weeks of Treatment
Description: The Sheehan Disability Scale (SDS) comprises self-rated items designed to measure impairment. The patient rates the extent to which his or her (1) work, (2) social life or leisure activities and (3) home life or family responsibilities are impaired on a 10-point visual analogue scales, on which 0 = normal functioning and 10 = severe functional impairment. The three items may be summed into a single dimensional measure of global functional impairment that ranges from 0 (unimpaired) to 30 (highly impaired). The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: SDS is a patient-reported outcome. The SDS Total Score is the sum of work, social life, or leisure activities, and home life or family responsibilities. FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 116 | 115 | 119 | 115 | 108
units on a scale | -6.11 (0.72) | -7.10 (0.74) | -6.52 (0.73) | -7.81 (0.74) | -7.91 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.6748, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-2.35 to 1.52], Standard Error of Mean 0.98 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.0871, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.70, 95% CI 2-sided [-3.64 to 0.25], Standard Error of Mean 0.99 — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.3186, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.99, 95% CI 2-sided [-2.94 to 0.96], Standard Error of Mean 0.99 — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0768, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.80, 95% CI 2-sided [-3.79 to 0.19], Standard Error of Mean 1.01 — No correction for multiplicity was made

7. Secondary Outcome: Proportion of Remitters at Week 8 (Remission Defined as a MADRS Total Score <=10)
Time Frame: Week 8
Population: FAS; LOCF; Logistic Regression
Measure: Number; unit: percentage of patients
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 155 | 151 | 149
percentage of patients | 33.8 | 32.9 | 36.1 | 35.8 | 34.9
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.6258, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 1.13, 95% CI 2-sided [0.70 to 1.81] — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.7178, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.68 to 1.76] — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.8651, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.59 to 1.55] — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.8563, Adjusting for Baseline — A nominal p-value is provided; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.65 to 1.69] — No correction for multiplicity was made

8. Secondary Outcome: Change From Baseline in HAM-A Total Score After 8 Weeks of Treatment
Description: The Hamilton Anxiety Rating Scale (HAM-A) consists of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behaviour at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic, and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total score from 0 to 56. The higher the score, the more severe.
Time Frame: Baseline and Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 154 | 155 | 151 | 148
units on a scale | -9.57 (0.63) | -9.87 (0.61) | -10.7 (0.61) | -10.6 (0.62) | -11.0 (0.62)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.1925, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.12, 95% CI 2-sided [-2.82 to 0.57], Standard Error of Mean 0.86 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.2434, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-2.72 to 0.69], Standard Error of Mean 0.87 — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.7246, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.30, 95% CI 2-sided [-2.00 to 1.39], Standard Error of Mean 0.86 — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.0981, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -1.45, 95% CI 2-sided [-3.16 to 0.27], Standard Error of Mean 0.87 — No correction for multiplicity was made

9. Secondary Outcome: Change From Baseline in CGI-S Score After 8 Weeks of Treatment
Description: The Clinical Global Impression - Severity of Illness (CGI-S) is a 7-point scale rated from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). The investigator should use his/her total clinical experience with this patient population to judge how mentally ill the patient is at the time of rating.
Time Frame: Baseline and Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 145 | 155 | 154 | 151 | 149
units on a scale | -1.64 (0.11) | -1.83 (0.10) | -1.81 (0.10) | -1.83 (0.10) | -1.82 (0.10)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.2285, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.46 to 0.11], Standard Error of Mean 0.14 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.1794, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.48 to 0.09], Standard Error of Mean 0.15 — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.1741, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.20, 95% CI 2-sided [-0.48 to 0.09], Standard Error of Mean 0.14 — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.2247, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.46 to 0.11], Standard Error of Mean 0.15 — No correction for multiplicity was made

10. Secondary Outcome: Change From Baseline in ASEX Total Score After 8 Weeks of Treatment
Description: The Arizona Sexual Experience Scale (ASEX) is a 5-item, patient self-rated scale that evaluates a patient's recent sexual experience. Patients are asked to assess their own experience over the last week (for example, "How strong is your sex drive?", "Are your orgasms satisfying?") and respond on a 6-point scale for each item. The ASEX is used to identify individuals with sexual dysfunction. Possible total score ranges from 5 to 30, with the higher score indicating more patient sexual dysfunction. A negative change indicates a lower sexual dysfunction.
Time Frame: Baseline and Week 8
Population: FAS; LOCF; ANCOVA
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 74 | 77 | 76 | 75 | 72
units on a scale | -0.41 (0.65) | -0.53 (0.62) | -0.66 (0.64) | -0.62 (0.62) | -0.38 (0.64)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.7789, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.24, 95% CI 2-sided [-1.93 to 1.45], Standard Error of Mean 0.86 — No correction for multiplicity was made
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.8121, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-1.91 to 1.50], Standard Error of Mean 0.87 — No correction for multiplicity was made
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.8918, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = -0.12, 95% CI 2-sided [-1.82 to 1.59], Standard Error of Mean 0.87 — No correction for multiplicity was made
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.9720, ANCOVA — A nominal p-value is provided; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-1.69 to 1.75], Standard Error of Mean 0.87 — No correction for multiplicity was made

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: 8-week double-blind treatment period and 4-week safety follow-up period Other Adverse Events: 8-week double-blind treatment period
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 3/148 | 1/155 | 3/157 | 2/151 | 2/155
Other Adverse Events (participants affected / at risk) | 64/148 | 61/155 | 63/157 | 62/151 | 93/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=148) | Vortioxetine 2.5 mg (N=155) | Vortioxetine 5 mg (N=157) | Vortioxetine 10 mg (N=151) | Duloxetine 60 mg (N=155)
Middle ear effusion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Serotonin syndrome (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Adenomyosis (Reproductive system and breast disorders) | 1/103 | 0/110 | 0/104 | 0/100 | 0/105
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=148) | Vortioxetine 2.5 mg (N=155) | Vortioxetine 5 mg (N=157) | Vortioxetine 10 mg (N=151) | Duloxetine 60 mg (N=155)
Constipation (Gastrointestinal disorders) | 6 | 3 | 5 | 3 | 10
Diarrhoea (Gastrointestinal disorders) | 10 | 7 | 3 | 8 | 7
Dry mouth (Gastrointestinal disorders) | 11 | 6 | 9 | 6 | 12
Nausea (Gastrointestinal disorders) | 13 | 26 | 26 | 33 | 52
Vomiting (Gastrointestinal disorders) | 5 | 6 | 6 | 7 | 11
Fatigue (General disorders) | 3 | 1 | 3 | 3 | 8
Nasopharyngitis (Infections and infestations) | 6 | 12 | 11 | 4 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 2 | 1 | 12
Dizziness (Nervous system disorders) | 10 | 7 | 5 | 6 | 25
Headache (Nervous system disorders) | 24 | 22 | 16 | 19 | 22
Somnolence (Nervous system disorders) | 5 | 5 | 4 | 5 | 11
Insomnia (Psychiatric disorders) | 6 | 8 | 11 | 3 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 4 | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The main publication has to be published before any sub-publications. H. Lundbeck A/S follows the Vancouver declaration with respect to authorship.